CLINICAL TRIAL: NCT05372640
Title: A Phase 1 Study of BET Bromodomain Inhibitor ZEN003694 in Combination With the CDK4/6 Inhibitor Abemaciclib in Patients With NUT Carcinoma, Breast Cancer and Other Solid Tumors
Brief Title: Testing the Safety and Efficacy of the Combination of Two Anti-cancer Drugs, ZEN003694 and Abemaciclib, for Adult and Pediatric Patients (12-17 Years) With Metastatic or Unresectable NUT Carcinoma, Breast Cancer and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-04100; NCI-2022-04100 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10509 (Other: Dana-Farber - Harvard Cancer Center LAO); 10509 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2022-05-12; First posted 2022-05-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Malignant Solid Neoplasm; Unresectable Breast Carcinoma; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — abemaciclib; Biopsy; Specimen Handling; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ZEN003694, abemaciclib) (Experimental): Patients receive ZEN003694 PO QD on days 1-28 or 5 days on and 2 days off of each cycle, and abemaciclib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo imaging evaluation, blood sample collection and tumor biopsy throughout the study.
  Interventions: Drug: Abemaciclib; Drug: BET Bromodomain Inhibitor ZEN-3694; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Diagnostic Imaging Testing

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY 2835219; LY-2835219; LY2835219; Verzenio
Drug: BET Bromodomain Inhibitor ZEN-3694 — Given PO
  Other Names: BETi ZEN-3694; ZEN 3694; ZEN-3694; ZEN003694
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Diagnostic Imaging Testing — Undergo imaging evaluation
  Other Names: Diagnostic Imaging; Medical Imaging

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of a ZEN003694 when given together with abemaciclib in treating patients with NUT carcinoma, breast cancer or other solid tumors that have spread from where it first started (primary site) to other places in the body (metastatic) or cannot be removed by surgery (unresectable). ZEN003694 is an inhibitor of a family of proteins called the bromodomain and extra-terminal (BET). It may prevent the growth of tumor cells that overproduce BET protein. Abemaciclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving ZEN003694 and abemaciclib may help shrink or stabilize cancer in patients with NUT carcinoma, breast cancer or other solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of the combination of BET bromodomain inhibitor ZEN-3694 (ZEN003694) and abemaciclib.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. Determine the preliminary rates of progression-free survival (PFS), overall survival (OS), overall response rate (ORR), time to response (TTR) and duration of response (DoR) for the combination of ZEN003694 and abemaciclib in participants utilizing Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

III. Evaluate the pharmacokinetic (PK) profile of the combination.

EXPLORATORY OBJECTIVE:

I. Explore potential biomarker indicators of response and resistance in tumor tissue and blood samples.

OUTLINE: This is a dose-escalation study of BET bromodomain inhibitor ZEN-3694 followed by a dose expansion study.

Patients receive ZEN003694 orally (PO) once daily (QD) on days 1-28 or 5 days on and 2 days off of each cycle, and abemaciclib PO twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo imaging evaluation, blood sample collection and tumor biopsy throughout the study.

After completion of study treatment, patients are followed up for 30 days, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Dose Escalation Cohort Only: Participants must have evaluable disease or measurable disease per RECIST 1.1 criteria
* Dose Expansion Cohort Only:

  * Participants must have a diagnosis of NUT carcinoma (NC) based on standard criteria for the disease, with diagnostic testing performed in a Clinical Laboratory Improvement Act (CLIA) certified laboratory:

    * Ectopic expression of NUT protein per World Health Organization (WHO) criteria as determined by immunohistochemistry (IHC) testing, OR
    * Detection of the NUT gene translocation as determined by fluorescence in situ hybridization (FISH) testing
    * Detection of the NUT gene translocation as determined by either deoxyribonucleic acid (DNA) next-generation sequencing (NGS) or ribonucleic acid (RNA) sequencing.
  * Participants must have measurable disease per RECIST 1.1 criteria
* Any number of prior lines of therapy in the metastatic setting are allowed, including prior BET inhibitor therapy and prior CDK4/6 inhibitor therapy
* Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] grade =< 1) from the acute effects of chemotherapy except for residual alopecia or grade 2 peripheral neuropathy
* Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy
* Participants may have previously undergone surgical resection
* Age >= 12 years. Patients 12-17 years of age must be > 40 kg at enrollment. Patients 12-17 years of age will not participate in the mandatory tumor biopsies. Since there is no data on patients less than 18 years of age, this population may require lower doses and additional safety precautions and should be closely monitored. Because no dosing or adverse event data are currently available on the use of ZEN003694 in combination with abemaciclib in patients <12 years of age, younger children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 for participants >= 16 years of age, Lansky >= 50% if < 16 years of age
* Hemoglobin >= 8 g/dL; Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 1 x 10^11/L
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) for age. Patients with Gilbert's syndrome with a total bilirubin =< 2.0 times ULN and direct bilirubin within normal limits are permitted
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN for age
* Serum or plasma creatinine =< 1.5 x institutional ULN OR calculated creatinine clearance >= 50 mL/min (via the chronic kidney disease epidemiology (CKD-EPI) glomerular filtration rate estimation for participants >= 18 years old, or 60 mL/min/1.73m^2 for patients 12-17 years as calculated based on bedside Schwartz formula)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load. Hepatitis C (HepC antibody) testing is required. Hepatitis C RNA is optional; however, a confirmatory negative Hepatitis C RNA test must be obtained to be able to enroll participants with positive Hepatitis C antibody due to prior resolved disease
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression and has been clinically stable for at least 1 month. Patients must meet the following criteria:

  * Disease outside the CNS is present
  * Recovery from acute toxicity associated with the treatment to =< CTCAE grade 1 or baseline (with the exception of alopecia), with no requirement for escalating doses of corticosteroids over the past 7 days
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients should be New York Heart Association Functional Classification of class 2B or better
* Ability to swallow and retain oral medications
* The effects of ZEN00364 and abemaciclib on the developing human fetus are unknown. For this reason and because BETi and CDKi-inhibiting agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Women of child-bearing potential must have a negative pregnancy test prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men and women treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 weeks after completion of ZEN003694 and abemaciclib administration

  * For female subjects of child-bearing potentially receiving ZEN003694, hormonal means of birth control alone, such as oral, injectable, dermal, subdermal or topical contraceptives are NOT acceptable forms of birth control given that their efficacy has not been evaluated when given in combination with the investigational drugs. "Adequate contraception" is defined as the following:

    * Contraceptive methods with a failure rate of =< 1% used in combination with the barrier method. The following contraceptive methods are acceptable to use in combination with the barrier method: intrauterine device (IUD), intrauterine system (IUS), or oral contraceptive pills (OCPs) that meet the < 1% failure rate as stated in the product label. Note: Hormonal IUDs/OCPs may only be used if the following criteria are met: male condoms are required AND subjects are informed of the potential for reduced systemic hormone levels from the IUD/OCP when taking ZEN003694. Alternatively, male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records
  * Male subjects with female partners of child-bearing potential must use one of the following contraceptive methods:

    * Vasectomy with documentation of azoospermia OR
    * Condom use PLUS partner use of a highly effective contraceptive (=< 1% rate of failure per year) such as intrauterine device or system, or hormonal birth control such as contraceptive subdermal implant, combined estrogen and progestogen oral contraceptive, injectable progestogen, contraceptive vaginal ring, or percutaneous contraceptive patches
  * Male subjects should not donate sperm while on study and for 12 weeks after the last dose of study medication. Male subjects whose partners are or become pregnant must continue to use condoms for 12 weeks after the last dose of study medication
* Women of childbearing potential must have a negative pregnancy test within 7 days of starting treatment
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity who have a legally-authorized representative (LAR) and/or family member available may be eligible after discussion with the Principal Investigator of this study. There will be a separate assent process for minors

Exclusion Criteria:

* Participants who have had cytotoxic chemotherapy, immunotherapy, or other investigational therapy within 2 weeks prior to entering the study. There is a two week required washout period for previous BET inhibitor therapy
* Participants who have had radiotherapy within at least 2 weeks prior to entering the study. Stereotactic radiosurgery (SRS) within 1 week prior to entering the study will be allowed
* Participants who have had major surgery within 3 weeks prior to entering the study
* Participants who have received tyrosine kinase inhibitors (TKIs) or small molecules within 5 half-lives or 1 week (whichever is shorter) of study entry
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ZEN003694 or abemaciclib
* Patients requiring medications or substances that are strong inhibitors or strong inducers of CYP3A4 or CYP3A enzymes are ineligible. Strong inhibitors or inducers of CYP3A4 must be discontinued at least 7 days prior to the first dose of ZEN003694 and abemaciclib. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness, including but not limited to: ongoing or active infection requiring systemic therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment (e.g. estimated creatinine clearance < 30ml/min), history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea that, in the judgment of the investigator, would preclude participation in this study
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 or substrates of CYP1A2 with narrow therapeutic windows are ineligible. Strong inhibitors or inducers of CYP3A4 must be discontinued at least 7 days prior to the first dose of ZEN003694. As proton pump inhibitors (PPIs), H2 receptor antagonists, and antacids may alter the pharmacokinetics of ZEN003694 by reducing ZEN003694 exposure, patients receiving proton pump inhibitors are ineligible. If H2 blockers or other acid reducing agents are used concomitantly with ZEN003694, a staggered dosing schedule should be used. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Pregnant women are excluded from this study because ZEN003694 is a BETi agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ZEN003694, breastfeeding should be discontinued if the mother is treated with ZEN003694. These potential risks may also apply to other agents used in this study
* Fridericia's correction formula (QTcF) >= 450 msec on screening electrocardiogram (ECG) (machine or manual read allowed). Patients should avoid medications which prolong the QT
* Patients receiving any medications or substances that are Factor Xa inhibitors (i.e., rivaroxaban, apixaban, betrixaban, edoxaban otamixaban, letaxaban, eribaxaban) or Factor IIa inhibitors (i.e., dabigatran). Low molecular weight heparin is allowed
* Patients with radiation to > 25% of the bone marrow
* Patients who have had a bone-targeted radionuclide within 6 weeks of the first dose of ZEN003694
* Myocardial infarction or unstable angina within 6 months prior to the first dose of ZEN003694
* Impairment of gastrointestinal function that may significantly alter the absorption of ZEN003694 and/or abemaciclib
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose or recommended phase 2 dose (Phase I dose escalation) | During the first cycle of therapy (28 days)
  The toxicity of the combination will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version (v). 5.0 criteria.
Incidence of adverse events (Phase I dose expansion) | Up to 5 years
  Safety will be reported with descriptive statistics. Toxicity will be graded according to National Cancer Institute CTCAE, v5.0. Toxicities will be summarized by maximum grade and by treatment arm. Incidence rate of each toxicity will be reported with 95% exact confidence intervals.
Overall response rate (Phase I dose expansion) | Up to 5 years
  Will be graded as complete response (CR), partial response (PR), stable disease (SD) and progressive disease.
Clinical benefit rate (CBR) (Phase I dose expansion) | Up to 5 years
  Clinical benefit is defined as CR, PR or SD >= 24 weeks according to Response Evaluation Criteria in Solid Tumors 1.1. CBR will be reported with 90% exact confidence intervals.
Duration of response (DoR) (Phase I dose expansion) | From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 5 years
  Median DOR will be reported with ranges.
Time to response (TTR) (Phase I dose expansion) | From the time initiation of therapy to the time measurement criteria are met for CR or PR (whichever is first recorded), assessed up to 5 years
  Median DOR will be reported with ranges.
Overall survival (Phase I dose expansion) | From study enrollment until death due to any cause, assessed up to 5 years
Progression free survival (Phase I dose expansion) | From study enrollment until the identification of disease progression or death, assessed up to 5 years

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | Up to 5 years
  Designed the PK sampling to enable simultaneous estimation of individual pharmacokinetic parameters of abemaciclib, ZEN003694, and their respective metabolites using nonlinear mixed effects modeling. Will compare the ratio of observed/historical 90% confidence interval of abemaciclib exposure.
Thymidine kinase (TK) | Up to 5 years
  Will compare exposures of abemaciclib and abemaciclib metabolites to TK activity at cycle 1 day 15 and beyond and also change in TK activity versus clinical outcomes.

OTHER OUTCOMES:
Analysis of ATAC-sequence data | Up to 5 years
  An internal pipeline will be used to perform quality control and data pre-processing. Burrows-Wheeler Aligner will be used for read mapping against the hg19 map using default parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Luo, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (7):
- United States (7):
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm